CLINICAL TRIAL: NCT05359393
Title: Radiotherapy Followed by Chemotherapy and Anti-PD-1 Immunotherapy in MSS Rectal Cancer With Resectable Liver/ Pulmonary Metastasis(Miracle-1): A Prospective, Single Arm, Multi-Center, Phase II Clinical Trial
Brief Title: A Combination Therapy Including Anti-PD-1 Immunotherapy in MSS Rectal Cancer With Resectable Distal Metastasis
Acronym: Miracle-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Miracle-1
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Advanced Rectal Cancer; Liver Metastasis; Pulmonary Metastasis; Microsatellite Stable Colorectal Carcinoma
MeSH Terms: interventions — Immunotherapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- resectable group (Experimental): In this group, we propose a combination therapy, preoperative short-course radiotherapy followed by neoadjuvant chemotherapy and anti-PD-1 immunotherapy, for microsatellite-stable patients with locally advanced rectal cancer and resectable liver/pulmonary metastasis.
  Interventions: Combination Product: a combination therapy including tislelizumab

INTERVENTIONS:
Combination Product: a combination therapy including tislelizumab — Patients will receive tislelizumab in combination with neoadjuvant radiotherapy and chemotherapy, and will be evaluated 2-3 weeks after completion of the treatment. Those patients who achieve complete clinical regression of the lesion can choose observation, but for those without CCR, surgical resection (TME of the primary lesion, surgical resection of metastases or other destructive local treatment) will be applied. Patients will continue to receive tislelizumab for one year after surgery or during observation.
  For liver/pulmonary metastasis, the treatment plan is to implement large fraction radiotherapy for 4-8 times. For primary rectum lesion, short-course radiotherapy regimen through intensity-modulated radiotherapy will be applied with dose of 25Gy/5Fx.
  Immunotherapy contains anti-PD-1 monoclonal antibody, Tislelizumab(200mg, d1, q3w x6, i.v). Chemotherapy adopts CAPEOX plan, including Capecitabine(1000mg/m2 bid, d1-14, p.o) and oxaliplatin(130mg/m2, d1, i.v).
  Other Names: preoperative radiotherapy combined with immunotherapy and chemotherapy

SUMMARY:
Although patients with locally advanced rectal cancer and resectable liver/pulmonary metastasis could benefit from surgery resection, these patients still have a poorer prognosis compared to those without distal metastasis. Based on previous studies, there is no confirmation of whether these patients could benefit from preoperative immunotherapy combined with conventional chemoradiotherapy. This study proposes a combination therapy, preoperative short-course radiotherapy followed by neoadjuvant chemotherapy and anti-PD-1 immunotherapy, for microsatellite-stable patients with locally advanced rectal cancer and resectable liver/pulmonary metastasis, to assess its impact on tumor retreat, decline of postoperative metastasis and recurrence, and the disease-free survival and overall survival of patients. Besides, this study will provide high-level medical evidence for future clinical treatment of patients with advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~75;
* Patient signs informed consent;
* ECOG score 0~1;
* Initial colonoscopy and pathology: adenocarcinoma;
* MRI: rectal cancer located less than 10cm from the anus;
* Imaging confirms that there are measurable metastases in the liver or lung, which are evaluated as NED acceptable by MDT discussion;
* no previous treatment;
* Patients have adequate organ function;
* No contraindications to surgery or chemoradiation;
* The relevant test results within 7 days before the first dose must meet the following requirements:

  1. Blood routine examination (no blood transfusion within 7 days before screening, no correction with hematopoietic stimulating factor drugs):

     * Hb≥90g/L
     * ANC≥1.5×10^9/L; LC≥0.5×10^9/L;
     * PLT≥100×10^9/L;
     * WBC≥3.0×10^9/L, ≤15×10^9/L;
  2. Blood chemistry (no blood transfusion or albumin within 7 days prior to screening):

     * ALT, AST≤1.5 ULN;
     * ALP≤2.5 ULN;
     * TBIL≤1.5 ULN;
     * Cr≤1.5 ULN, CrCL≥50 mL/min;
     * PT, APTT≤1.5 ULN, INR≤1.5 ULN(not receiving anticoagulation);
  3. TSH is within the normal range; if TSH is out of the normal range, FT3 and FT4 should be investigated. If the test results of FT3/FT4 cannot be obtained, T3 and T4 can be accepted. If the level of T3/T4 is normal, the patients can be selected.
  4. Urine test: urine protein<2+; if the urine protein≥2+, the 24-hour urine protein quantification must be≤1g;
  5. Echocardiography: LVEF≥55%;
  6. 12-lead ECG: Fridericia corrected QTcF<470 msec.
* Expected survival time >6 months;
* The gene status of KRAS, NRAS, BRAF and HER2 is clear;
* Patients with microsatellite stability or mismatch repair protein defects;
* Patients are willing and able to follow the protocol during the study, including receiving treatment and scheduled follow-up and examination.

Exclusion Criteria:

Patients will not be accepted into this study if they meet any of the following criteria:

1. History of tumor-related disease and treatment:

1. Age <18 or >75 years;
2. other malignancy within 5 years, except adequately treated carcinoma in situ of the cervix or squamous cell carcinoma of the skin, or largely controlled basal cell carcinoma of the skin;
3. malignant pleural effusion or malignant ascites;
4. patients with severe medical comorbidities that preclude radiotherapy and surgery;
5. previously treated;
6. clinical or radiological evidence of spinal cord compression or a tumor within 3mm of the spinal cord on MRI
7. the presence of distant metastases besides the liver and lungs, including brain, bone, ovarian, peritoneal and retroperitoneal multiple lymph node metastases;
8. Patients who are considered suitable for using intense systemic treatment to achieve conversion after MDT discussion;
9. pathological diagnosis of indolent cell carcinoma;
10. patients with microsatellite instability or dMMR;
11. patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. that require emergency surgical resection;

2. Co-morbidities and treatment history:

1. Presence of immunodeficiency disorders, including primary immunodeficiency disorders (e.g. caused by genetic factors) or secondary immunodeficiency disorders (e.g. caused by HIV infection or treatment related to immunological agents, etc.);
2. Presence of any autoimmune disease that still requires treatment or a previous history of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, rheumatic heart valve disease, glomerulonephritis, etc. Excluding hypothyroidism due to autoimmune thyroiditis requiring only hormone replacement therapy and type I diabetes with manageable and stable blood glucose;
3. known or suspected interstitial pneumonia; other moderate to severe lung disease that may interfere with the detection or management of drug-related pulmonary toxicity and severely affect respiratory function, including idiopathic pulmonary tissue fibrosis, mechanized pneumonia/occlusive fine bronchitis, etc.;
4. severe cardiovascular disease, including but not limited to conditions meeting NYHA criteria (Class III or higher), or myocardial infarction or cerebrovascular accident (cerebral ischaemia, symptomatic cerebral infarction, etc.) occurring within 3 months prior to the first dose, or unstable arrhythmia or unstable angina pectoris with coronary artery disease occurring within 1 month prior to the first dose, or congestive heart failure, or pre-existing symptomatic superior vena cava syndrome, etc.;
5. an arteriovenous thrombotic event, such as deep vein thrombosis and pulmonary embolism, within the previous 3 months;
6. history of live attenuated vaccination within 28 days prior to the first study dose or anticipated need for live attenuated vaccination during the study;
7. active hepatitis B (defined as positive hepatitis B virus surface antigen [HBsAg] test result and HBV-DNA test value ≥ 500 IU/ml);
8. Hepatitis C (defined as a positive test result for hepatitis C virus antibody [HCV-Ab]) ;
9. history of tuberculosis infection or treatment within 1 year prior to signing informed consent;
10. presence of severe infection within 4 weeks prior to first dose, including but not limited to bacteremia requiring hospitalization, severe pneumonia, etc.; or active infection requiring systemic antibiotic therapy according to NCI-CTCAE v5.0 grade ≥ 2 within 2 weeks prior to first dose, or unexplained fever >38.5°C during screening/prior to first dose (at the investigator's discretion, due to oncologic causes fever due to tumor causes may be enrolled);
11. previous allogeneic bone marrow transplantation or solid organ transplantation received or intended to be received;
12. Hemoptysis with a maximum daily hemoptysis of approximately ≥2.5 ml within 2 months prior to signing informed consent; clinically significant bleeding symptoms or a clear bleeding tendency within 1 month prior to signing informed consent, e.g. gastrointestinal bleeding, bleeding gastric ulcer, fecal occult blood ++ at baseline, vasculitis; known hereditary or acquired bleeding and thrombotic tendencies, e.g. hemophilia, impaired coagulation skills, thrombocytopenia, hypersplenism, etc.;
13. abnormal coagulation (INR > 1.5 or APTT > 1.5 × ULN) with bleeding tendency or undergoing thrombolysis or requiring long-term anticoagulation with warfarin or heparin, or requiring long-term antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day)
14. peripheral neuropathy ≥ grade 2 according to NCI-CTCAE v5.0;
15. Co-morbidities of other infectious diseases that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
NED rate | 1 years after treatment
  rate of no evidence of disease for one year

SECONDARY OUTCOMES:
Overall Survival | 5 years after surgery
  For patients who still survive when the final analysis takes place, the date of the last 1 contact will be recorded.
Disease Free Survival | 5 years after surgery
  DFS refers to the period of time between the date of surgery and the day of the patient's tumor recurrence or death (earliest occurrence).
Local Recurrence | 5 years after surgery
  The date of recurrence is defined as the date on which an objective examination yields a positive result.
Objective Response Rate | 5 years after surgery
  Percentage of patients with objective response to primary or metastatic lesions
Tumor Regression Rate | 5 years after surgery
  Surgical excision specimens are taken every 1 cm, and the sections are given to at least 2 pathologists for independent scoring
Acute toxicity associated with immunotherapy | from the beginning of treatment to 90 days after the end of immunotherapy
  According to the NCI CTCAE v5.0 assessment, the proportion of patients with treatment-related acute toxicity developed from the beginning of treatment to 90 days after the end of immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China